CLINICAL TRIAL: NCT01417169
Title: Efficacy and Safety in Micafungin Sodium for Prophylaxis Against Invasive Fungal Disease During Neutropenia in Pediatric & Adolescent Patients Undergoing Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Micafungin Prevention Study for Invasive Fungal Disease in Pediatric & Adolescent Patients Undergoing Autologous Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SNUCH-1102
Record Dates: First submitted 2011-08-09; First posted 2011-08-16 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Neutropenia; Fungal Disease
MeSH Terms: conditions — Neutropenia; Mycoses | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Micafungin (Experimental)
  Interventions: Drug: micafungin

INTERVENTIONS:
Drug: micafungin — Eligible patients who provided informed consent form will be administered micafungin at 50 mg/day (1mg/kg/day for patients weighting <50kg) as 1-h infusion. Infusion of Micafungin will be started on the day -2 of the conditioning course of autologous stem cell transplantation
  Other Names: Micafungin sodium; Mycamine

SUMMARY:
This study is to evaluate safety and prophylaxis effect of micafungin after hematopoietic stem cell transplantation. Micafungin is administered until confirmation of neutrophil engraftment or treatment failure.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate absence of proven, probable, possible, suspected invasive fungal disease (IFDs) through the end of prophylaxis therapy and during 4 weeks after stopping of micafungin prophylaxis after Autologous hematopoietic stem cell transplantation in pediatric and adolescent neutropenia patients. Patients will receive micafungin until the earliest of the following: 1) neutrophil engraftment; 2) development of proven, provable, possible or suspected invasive fungal disease; 3) development of unacceptable drug toxicity; 4) withdrawal from study participation or discontinuation of study treatment. Safety profile of micafungin is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will receive autologous hematopoietic stem cell transplantation including 2nd autologous transplantation
2. Under 21 years old, pediatric, adolescent patients.

Exclusion Criteria:

1. Aspartate transaminase or alanine transaminase level > 5 times UNL
2. Bilirubin > 2.5 times UNL
3. History of allergy, sensitivity, or any serious reaction to an echinocandin
4. Invasive fungal disease at the time of enrolment
5. Systemic antifungal therapy within 72 hrs before administration of the first dose of study drug
6. Positive pregnancy test

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Absence rate of IFDs assessed by physical examination and serum galactomannan test | 4 weeks
  Absence of proven, probable, possible invasive fungal disease (IFDs) through the end of prophylaxis therapy and during 4 weeks after stopping of Micafungin prophyalxis after HSCT

SECONDARY OUTCOMES:
Survival rate | 100 days
  IFD-related mortality
Safety assessed by lab-test and adverse events | 4 weeks
  Safety profiles

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, M.D, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea